CLINICAL TRIAL: NCT02177357
Title: Pramipexole: Efficacy, Safety and Tolerability Study in Untreated and Levodopa-Treated Parkinson's Disease Patients, a Multinational Study
Brief Title: Pramipexole in Untreated and Levodopa-treated Parkinson's Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 248.362
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

ARMS (2):
- Pramipexole - escalation dose (Experimental)
  Interventions: Drug: Pramipexole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pramipexole
  Arms: Pramipexole - escalation dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objectives of this study were to evaluate the efficacy, safety, and tolerability of pramipexole, as single-agent therapy or in combination with levodopa, in patients with Parkinson disease living in Hong Kong and Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 30 years of age with a diagnosis of symptomatic, idiopathic Parkinson disease, stage 1-4 on the Modified Hoehn and Yahr Scale
* Females either surgically sterile or at least 2 years postmenopausal, or using a reliable method of contraception for at least 2 months prior to study entry
* Females of childbearing potential with a negative pregnancy test at the screening visit and not nursing
* Patients with at least 3 of the 4 cardinal signs of Parkinson disease (i.e., rigidity, bradykinesia, resting tremor, postural instability) and without any other known or Suspected cause for their Parkinsonism
* Patients on levodopa therapy who show a good response to levodopa and be on a stable dosage of levodopa for least 1 month prior to study entry
* Patients able to take oral medication
* Patients must give voluntary written consent for study participation and must sign a Patient Informed Consent Form at the screening visit, prior to initiation of any study-related procedures

Exclusion Criteria:

* Atypical parkinsonian syndromes secondary to drugs (e.g., metoclopramide, flunarizine), metabolic disorders (e.g., Wilson disease), encephalitis, or degenerative diseases (e.g., progressive supranuclear palsy, multiple-system atrophy)
* Dementia that could impair compliance with medication and/or preclude giving informed consent (i.e., Mini-Mental Status Examination score ≤22)
* History of psychosis
* History of active epilepsy (e.g., occurrence of a seizure) within 1 year prior to screening
* Second or third degree atrioventricular block or sick sinus syndrome, resting heart rate below 50 beats per minute, congestive heart failure (New York Heart Association functional Class III or IV), myocardial infarction within 6 months of randomization, or other clinically significant heart conditions (e.g., coronary artery disease) that might negatively affect the possibility of the patient completing the study
* Clinically significant liver disease that may prevent the patient from completing the study and/or elevation in total bilirubin, alkaline phosphatase, lactate dehydrogenase (LDH), serum glutamate pyruvate transaminase (SGPT), or serum glutamate oxaloacetate transaminase (SGOT) of >1.5 times the upper limit of the normal values
* Clinically significant renal disease that may prevent the patient from completing the study and/or elevation in serum creatinine of >1.5 times the upper limit of the normal values
* Presence of active neoplastic disease
* Surgery within 6 months of the baseline/randomization visit which, in the opinion of the investigator, might negatively impact the patient's participation in the study, or any history of stereotaxic brain surgery (e.g., thalamotomy, pallidotomy, or any other deep brain stimulation for reduction of parkinsonian symptoms)
* Supine systolic blood pressure less than 100 mm Hg or evidence of a ≥20-mm Hg decline in systolic blood pressure at 2 minutes after standing, compared with the previous supine systolic blood pressure obtained after 5 minutes of quiet rest, if the decline in blood pressure upon standing is associated with symptoms (i.e., symptomatic orthostatic hypotension)
* Use of dopamine agonist medications (e.g., bromocriptine, pergolide) in the 2 months prior to study entry (allowed medications: selegiline, anticholinergics, and amantadine therapy at a stable dosage for 60 days prior to study entry and remaining stable throughout the study)
* Use of neuroleptics, alpha-methyldopa, or flunarizine within the past 6 months
* Use of any of the following drugs within 3 months of study entry: methylphenidate, cinnarizine, reserpine, amphetamine, and monoamine oxidase-A inhibitors (e.g., pargyline, phenelzine, or tranylcypromine)
* Use of pramipexole within the past 3 months or a history of adverse reaction or allergy to pramipexole
* Unstable dosage of centrally active therapies (e.g., hypnotics, antidepressants, anxiolytics) within the past 60 days
* Electroconvulsive therapy within 90 days of the baseline/randomization visit
* Participation in other investigational drug studies or receipt of other investigational drugs within 30 days prior to baseline/randomization. Investigational drugs for Parkinson disease must have been discontinued for 90 days prior to baseline/randomization. Additionally, patients previously randomized into this study and who then discontinued study participation are not to be re-entered into the study
* Positive hepatitis B screen (assessed at the screening visit)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 1998-11; Primary Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the sum of the UPDRS (Unified Parkinson Disease Rating Scale) Parts II and III total scores. | up to 15 weeks
Number of patients with clinically significant changes in vital signs | up to 15 weeks
Number of patients with abnormal changes in laboratory parameters | up to 15 weeks
Number of patients with abnormal changes in 12-lead ECG (electrocardiogram) | up to 15 weeks
Number of patients with adverse events | up to 15 weeks

SECONDARY OUTCOMES:
Change from baseline in the individual UPDRS Part II and Part III total scores | up to 15 weeks
Change from baseline the individual items in the UPDRS Part II and Part III | up to 15 weeks
Change from baseline in the Modified Hoehn and Yahr Scale | up to 15 weeks
Change from baseline in the number of "off" hours in those patients who had been on levodopa therapy | up to 15 weeks
Change from baseline in the Mini-Mental Status Examination | up to 15 weeks